CLINICAL TRIAL: NCT02959970
Title: An Open-Label Phase 4 Safety and Efficacy Trial of ACZONE (Dapsone) Gel, 7.5% in 9 to 11 Year-Old Patients With Acne Vulgaris
Brief Title: Safety and Efficacy Trial of ACZONE (Dapsone) Gel, 7.5% in 9 to 11 Year-Old Patients With Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1679-401-006
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PK Cohort: ACZONE 7.5% (Experimental): Participants applied ACZONE 7.5 % gel topically, once-daily to the entire face, neck, upper chest, upper back and shoulders starting from Day 1 under maximal use conditions (2 grams per day) for Day 8 consecutive days, followed by a thin layer to their face and acne-affected areas on the upper chest, upper back, and shoulders for next 11 weeks.
  Interventions: Drug: dapsone gel
- Non-PK Cohort: ACZONE 7.5% (Experimental): Participants applied ACZONE 7.5% gel topically, once-daily in a thin layer to their face and acne-affected areas on upper chest, upper back, and shoulders for 12 weeks.
  Interventions: Drug: dapsone gel

INTERVENTIONS:
Drug: dapsone gel — Dapsone (ACZONE) 7.5% gel topically once daily.
  Other Names: ACZONE

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK) and efficacy of ACZONE Gel, 7.5% administered topically once-daily for 12 weeks in 9 to 11 year-olds with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

-Has acne vulgaris on the face, including the nose, with 20 to 100 total lesions (noninflammatory and/or inflammatory).

Exclusion Criteria:

* Has uncontrolled systemic disease(s)
* Has severe cystic acne, acne conglobata, acne fulminans, or secondary acne (chloracne, drug-induced acne)
* Has used topical dapsone within 1 month prior to the screening
* Has used oral dapsone within 2 months prior to screening.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Truong, Study Director — Allergan
Locations (20):
- United States (20):
  - Kirklin Clinic, Birmingham, Alabama
  - Center for Dermatology Clinical Research, Fremont, California
  - Quest Dermatology Research, Northridge, California
  - Southern California Dermatology, Santa Ana, California
  - Redwood Family Dermatology, Santa Rosa, California
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Baumann Cosmetic and Research Institute, Miami Beach, Florida
  - Dermresearch, PLLC, Louisville, Kentucky
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Saint Louis University Dermatology, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Skin Specialty Dermatology, New York, New York
  - Health Sciences/Department of Dermatology, Winston-Salem, North Carolina
  - KGL Skin Study Center, Broomall, Pennsylvania
  - Department of Dermatology, UPCII, Hershey, Pennsylvania
  - Arlington Research Center, Inc., Arlington, Texas
  - DermResearch, LLC, Austin, Texas
  - University of Texas Medical School at Houston, Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Premier Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 sites in United States (US) between 31 October 2016 (first participant first visit) and 09 March 2018 (last participant last visit).
Pre-assignment Details: A total of 105 participants were screened, out of which 100 participants were enrolled into either of the 2 cohorts, Pharmacokinetic (PK) Cohort and Non-PK Cohort.
Period: Overall Study
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Started | 17 | 83
Completed | 15 | 76
Not Completed | 2 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one application of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5% | Total
Number analyzed (Participants) | 17 | 83 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (0.9) | 10.4 (0.7) | 10.4 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 59 | 74
  Male | 2 | 24 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 23 | 26
  Not Hispanic or Latino | 14 | 60 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 9 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 19 | 24
  White | 9 | 53 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE was defined as "any untoward medical occurrence in a clinical trial participant (regardless of the administration of the study drug and its causal relationship to it). An AE could therefore, be any unfavorable and unintended medical occurrence during the participant's participation in the trial, including deterioration of a pre-existing medical condition, an abnormal clinically significant finding in a laboratory assessment, or an abnormal clinically significant finding in the physical examination or vital sign.
Time Frame: From Baseline (Day 1) until Week 12
Population: Safety population included all participants who received at least one application of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
Participants | 5 | 16

2. Primary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure
Description: Change from baseline in systolic and diastolic blood pressure was evaluated. Change from baseline was calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: Safety population included all participants who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Groups:
- Non-PK Cohort: ACZONE 7.5%: Participants applied ACZONE 7.5% gel topically, once-daily in a thin layer to the their face and acne-affected areas on upper chest, upper back, and shoulders for 12 weeks.
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
millimeter of mercury (mmHg)
  Systolic Blood Pressure | 3.9 (8.2) | 0.1 (10.1)
  Diastolic Blood Pressure | 2.3 (5.9) | 0.4 (9.1)

3. Primary Outcome: Change From Baseline in Heart Rate
Description: Change from baseline in heart rate was evaluated. Change from baseline was calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: Safety population included all participants who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
beats per minute (beats/min) | -0.8 (14.0) | 0.6 (9.5)

4. Primary Outcome: Change From Baseline in Respiratory Rate
Description: Change from baseline in respiratory rate was assessed. Change from baseline was calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: Safety population included all participants who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: breaths per minute (breaths/min)
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
breaths per minute (breaths/min) | 0.5 (2.4) | -0.1 (1.6)

5. Primary Outcome: Change From Baseline in Body Temperature
Description: Change from baseline in body temperature was assessed. Change from baseline was calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: Safety population included all participants who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: degree celsius (°C)
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
degree celsius (°C) | 0.08 (0.26) | 0.10 (0.38)

6. Primary Outcome: Change From Baseline in Weight
Description: Change from baseline in weight was assessed. Change from baseline was calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: Safety population included all participants who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
kilogram (kg) | 0.70 (1.98) | 1.48 (1.72)

7. Primary Outcome: Change From Baseline in Height
Description: Change from baseline in height was assessed. Change from baseline was calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: Safety population included all participants who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
centimeter (cm) | 0.21 (0.76) | 1.01 (1.77)

8. Primary Outcome: Local Dermal Tolerability: Number of Participants With Dryness, Scaling and Erythema as Assessed by Investigator
Description: Local dermal tolerability was evaluated by investigator in terms of presence and absence of dryness, scaling and erythema symptoms and its severity in the areas of body where medication was applied. These symptoms were assessed by using a 4 - point scale of 0 - 3, where 0 = none (no dryness, scaling and erythema) and 3 = severe (marked roughness, heavy scale production and intense redness). The higher score indicated severe symptoms.
Time Frame: Week 12
Population: Safety population included all participants who received at least one application of study drug. Here, "number analyzed" signifies number of participants with available data for the specified category.
Measure: Number; unit: participants
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
participants
  Dryness: None (0): number analyzed (Participants) | 15 | 77
  Dryness: None (0) | 15 | 71
  Dryness: Mild (1): number analyzed (Participants) | 15 | 77
  Dryness: Mild (1) | 0 | 6
  Dryness: Moderate (2): number analyzed (Participants) | 15 | 77
  Dryness: Moderate (2) | 0 | 0
  Dryness: Severe (3): number analyzed (Participants) | 15 | 77
  Dryness: Severe (3) | 0 | 0
  Scaling: None (0): number analyzed (Participants) | 15 | 77
  Scaling: None (0) | 15 | 70
  Scaling: Mild (1): number analyzed (Participants) | 15 | 77
  Scaling: Mild (1) | 0 | 6
  Scaling: Moderate (2): number analyzed (Participants) | 15 | 77
  Scaling: Moderate (2) | 0 | 1
  Scaling: Severe (3): number analyzed (Participants) | 15 | 77
  Scaling: Severe (3) | 0 | 0
  Erythema: None (0): number analyzed (Participants) | 15 | 77
  Erythema: None (0) | 13 | 65
  Erythema: Mild (1): number analyzed (Participants) | 15 | 77
  Erythema: Mild (1) | 2 | 12
  Erythema: Moderate (2): number analyzed (Participants) | 15 | 77
  Erythema: Moderate (2) | 0 | 0
  Erythema: Severe (3): number analyzed (Participants) | 15 | 77
  Erythema: Severe (3) | 0 | 0

9. Primary Outcome: Local Dermal Tolerability: Number of Participants With Stinging/Burning Symptoms as Assessed by Participants
Description: Local dermal tolerability was evaluated by participants in terms of presence and absence of prickling pain sensation immediately after (within 5 minutes of dosing) and its severity in the areas of body where medication was applied (face). Stinging/burning symptoms were graded on a 4-point scale of 0 - 3 where 0 = none (no stinging/burning), 1 = mild (slight warm, tingling/stinging sensation; not really bothersome), 2 = moderate (definite warm, tingling/stinging sensation that is somewhat bothersome), 3 = severe (hot, tingling/stinging sensation that has caused definite discomfort). The higher score indicated severe symptoms.
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | PK Cohort: ACZONE 7.5% | Non-PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 17 | 83
participants
  None (0): number analyzed (Participants) | 15 | 77
  None (0) | 15 | 75
  Mild (1): number analyzed (Participants) | 15 | 77
  Mild (1) | 0 | 2
  Moderate (2): number analyzed (Participants) | 15 | 77
  Moderate (2) | 0 | 0
  Severe (3): number analyzed (Participants) | 15 | 77
  Severe (3) | 0 | 0

10. Other Pre Specified Outcome: Peak Plasma Concentration of Dapsone,Dapsone Hydroxylamine and N-acetyl Dapsone at Week 1
Description: The mean plasma peak (10 hours postdose) concentrations of dapsone, dapsone hydroxylamine and N-acetyl dapsone were reported.
Time Frame: Week 1 (Pre-dose and 10 hours post-dose)
Population: Pharmacokinetic (PK) population included all participants who received applications of study drug for at least 8 days under maximal use conditions and had evaluable blood samples for PK analysis.
Measure: Mean (Standard Deviation); unit: nanogram per milliter (ng/mL)
Arm/Group | PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 16
nanogram per milliter (ng/mL)
  Dapsone | 20.0 (12.5)
  Dapsone hydroxylamine | 1.40 (1.10)
  N-acetyl dapsone | 9.01 (7.37)

11. Other Pre Specified Outcome: Trough Plasma Concentration of Dapsone, Dapsone Hydroxylamine and N-acetyl Dapsone at Week 1
Description: The trough plasma concentrations of Dapsone, Dapsone hydroxylamine and N-acetyl dapsone were reported.
Time Frame: Week 1 (Pre-dose)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PK Cohort: ACZONE 7.5%
Number analyzed (Participants) | 16
ng/mL
  Dapsone | 17.2 (14.0)
  Dapsone hydroxylamine | 1.05 (0.979)
  N-acetyl dapsone | 7.02 (5.28)

12. Other Pre Specified Outcome: Absolute Change From Baseline in Inflammatory Lesion Counts
Description: Inflammatory lesion counts were the sum of counts of the following lesion types (face only): Papule - a small, red, solid elevation less than (<) 1.0 centimeter (cm) in diameter; Pustule - a small, circumscribed elevation of the skin that contains yellow-white exudate; Nodule - a circumscribed, elevated, solid lesion generally more than 1.0 cm in diameter with palpable depth; Cyst - a smooth, dome-shaped, elevated, freely moveable, skin-colored, round to ovoid lesion greater than 0.7 cm in diameter. Change from baseline was calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: Modified intent-to-treat (mITT) population included all enrolled participants who had a baseline assessment and at least one post-baseline assessment. This population was presented as combined data from both cohorts (PK Cohort: ACZONE 7.5% and Non-PK Cohort: ACZONE 7.5%).
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- ACZONE 7.5%: Participants applied ACZONE 7.5% gel topically, once-daily to their face for 12 weeks.
Arm/Group | ACZONE 7.5%
Number analyzed (Participants) | 98
lesions | -6.2 (9.3)

13. Other Pre Specified Outcome: Percent Change From Baseline in Inflammatory Lesion Counts
Description: Inflammatory lesion counts were the sum of counts of the following lesion types (face only): Papule - a small, red, solid elevation less than 1.0 cm in diameter; Pustule - a small, circumscribed elevation of the skin that contains yellow-white exudate; Nodule - a circumscribed, elevated, solid lesion generally more than 1.0 cm in diameter with palpable depth; Cyst - a smooth, dome-shaped, elevated, freely moveable, skin colored, round to ovoid lesion greater than 0.7 cm in diameter.
Time Frame: Baseline (Day 1), Week 12
Population: Modified intent-to-treat (mITT) population included all enrolled participants who had a baseline assessment and at least one post-baseline assessment.This population was presented as combined data from both cohorts (PK Cohort: ACZONE 7.5% and Non-PK Cohort: ACZONE 7.5%).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ACZONE 7.5%
Number analyzed (Participants) | 98
percent change | -56.38 (43.43)

14. Other Pre Specified Outcome: Absolute Change From Baseline in Non-inflammatory Lesion Counts
Description: Non-inflammatory lesion counts were defined as the sum of counts of the following lesion type (face only): open comedone - a pigmented dilated pilosebaceous orifice (blackhead); closed comedone - a tiny white papule (whitehead). Change from baseline was be calculated by subtracting post-dose value from the baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | ACZONE 7.5%
Number analyzed (Participants) | 98
lesions | -17.8 (17.0)

15. Other Pre Specified Outcome: Percent Change From Baseline in Non-inflammatory Lesion Counts
Description: Noninflammatory lesion counts were defined as the sum of counts of the following lesion type (face only): open comedone - a pigmented dilated pilosebaceous orifice (blackhead); closed comedone - a tiny white papule (whitehead).
Time Frame: Baseline (Day 1), Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ACZONE 7.5%
Number analyzed (Participants) | 98
percent change | -46.45 (69.90)

16. Other Pre Specified Outcome: Absolute Change From Baseline in Total Lesion Counts on Face
Description: Total lesion counts were defined as the sum of inflammatory lesion counts and noninflammatory lesion counts (face only). Change from baseline was be calculated by subtracting post-dose value from the baseline value.
Time Frame: Baseline (Day 1), Week 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | ACZONE 7.5%
Number analyzed (Participants) | 98
lesions | -24.0 (23.0)

17. Other Pre Specified Outcome: Percent Change From Baseline in Total Lesion Counts on Face
Description: Total lesion counts were defined as the sum of inflammatory lesion counts and noninflammatory lesion counts (face only).
Time Frame: Baseline (Day 1), Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ACZONE 7.5%
Number analyzed (Participants) | 98
percent change | -51.91 (33.53)

18. Other Pre Specified Outcome: Percentage of Participants With None (0) or Minimal (1) Score on the Investigator's Global Assessment (IGA) for Face
Description: Overall severity of acne vulgaris was evaluated by using a 5-point IGA scale: Clear (0) - (no comedones; papules or pustules, residual hyperpigmentation and erythema may be present); Almost clear (1) - (rare comedones; no more than a few small papules and pustules); Mild (2) - (easily recognizable comedones in limited numbers; +/- presence of small papules and pustules); Moderate (3) - (many comedones; +/- easily recognizable small and medium-sized papules; no nodules or cysts; Severe (4) - (widespread and numerous comedones; many small, medium-sized and large papules and pustules; nodules or cysts may or may not be present).
Time Frame: Week 12
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | ACZONE 7.5%
Number analyzed (Participants) | 98
percentage of participants | 46.7

19. Other Pre Specified Outcome: Percentage of Participants With None (0) or Minimal (1) Score Plus at Least a 2-Grade Improvement on the Investigator's Global Assessment (IGA) for Face
Description: as for outcome 18
Time Frame: Week 12
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | ACZONE 7.5%
Number analyzed (Participants) | 98
percentage of participants | 19.6

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) until Week 12
Description: Reported AEs were treatment-emergent AEs that developed/worsened during the 'on-treatment period' (defined as the period from the time of the first dose of the drug until 12 weeks). The analysis was performed on the safety population.
Groups:
- PK Cohort: Participants applied ACZONE 7.5 % gel topically, once-daily to the entire face, neck, upper chest, upper back and shoulders starting from Day 1 under maximal use conditions (2 grams per day) for Day 8 consecutive days, followed by a thin layer to their face and acne-affected areas on the upper chest, upper back, and shoulders for next 11 weeks.
- Non-PK Cohort: Participants applied ACZONE 7.5% gel topically, once-daily in a thin layer to their face and acne-affected areas on upper chest, upper back, and shoulders for 12 weeks.
Arm/Group | PK Cohort | Non-PK Cohort
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/83
Other Adverse Events (participants affected / at risk) | 5/17 | 16/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PK Cohort (N=17) | Non-PK Cohort (N=83)
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2
Pharyngitis streptococcal (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 1 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Blood iron decreased (Investigations) | 0 | 1
Vitamin D decreased (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin pigmentation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship and manuscript composition will reflect joint cooperation between multiple investigators and sites and the Sponsor's personnel. Authorship will be established prior to the writing of the manuscript. As this study involves multiple centers, no individual publications will be allowed prior to completion of the final report of the multicenter study except as agreed with the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT02959970/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT02959970/SAP_001.pdf